CLINICAL TRIAL: NCT01918813
Title: Risk of Methicillin-resistant S.Aureus (MRSA) Infections in MRSA Carrier Under Introduction of Rapid MRSA Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chikara Tashiro (Other)
Responsible Party: Sponsor-Investigator, Chikara Tashiro, Director of hospital, Hyogo Medical University
Organization: Hyogo Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Hyogo college of Medicine 749
Record Dates: First submitted 2013-08-05; First posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Inflammatory Bowel Disease; Hepatobiliary Disease; Pancreas Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Digestive System Diseases; Pancreatic Diseases | interventions — Vancomycin; Mupirocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preoperative MRSA nasal colonization (Experimental): Interventions in arm of preoperative MRSA nasal colonization consisted of antibiotic prophylaxis with a single dose of vancomycin 1g in addition to cephalosporins, and topical decolonization of MRSA with application of 2% mupirocin ointment twice daily to nares for 5 days
  Interventions: Drug: vancomycin, mupirocin ointment

INTERVENTIONS:
Drug: vancomycin, mupirocin ointment — contact precautions, topical decolonization of MRSA by a bath with 4% chlorhexidine daily for 3-5 days
  Other Names: vancomycin, bactroban ointment

SUMMARY:
This study was designed to evaluate the effect of a targeted preoperative Methicillin-resistant Staphylococcus aureus (MRSA) detection by polymerase chain reaction (PCR) on either endogenous or exogenous postoperative MRSA infections in a high risk population undergoing gastroenterological surgery. The primary endpoint was to investigate whether the potentially high incidence of MRSA infections in patients with MRSA nasal colonization before surgery can be prevented with a PCR-based strategy. The second endpoint was to investigate the impact of acquisition of MRSA colonization after surgery on the occurrence of MRSA infections. Investigators hypothesize that postoperative MRSA infection is prevented by a targeted screening strategy in preoperative MRSA carrier, and there is limited effect in patients with postoperative MRSA acquisition.

DETAILED DESCRIPTION:
Target screening for nasal carriage of MRSA by polymerase chain reaction (PCR) was performed before or on admission. In order to identify MRSA nasal acquisition while on the ward, all patients who were negative before surgery were re-screened every 7 days until discharge. The inclusion criteria for screening were patients undergoing inflammatory bowel disease surgery on ward A, and those undergoing major hepato-biliary-pancreatic surgery on ward B. Investigators classified enrolled patients into preoperative MRSA nasal carriage, postoperative nasal acquisition in patients who were negative for PCR assay before surgery, and non-nasal MRSA carriage during hospitalization. Development of postoperative infections caused by MRSA was assessed according to the nasal MRSA carriage status. MRSA infections rate was also compared between the 2-years of the intervention period and the previous 2-year control period on each ward.

Control measures in identified MRSA carriers consisted of contact precautions, antibiotic prophylaxis with a single dose of vancomycin 1g in addition to cephalosporins, and topical decolonization of MRSA (application of 2% mupirocin ointment twice daily to nares for 5 days and a bath with 4% chlorhexidine daily for 3-5 days). Although contact precautions were used when caring for MRSA-colonized patients, isolation/cohorting was not routinely practiced.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing inflammatory bowel disease (IBD) surgery
* patients undergoing major hepato-biliary-pancreatic surgery

Exclusion Criteria:

* emergency surgery,
* age less than 18 years old
* known allergy to mupirocin or chlorhexidine.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 662 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The incidence of MRSA infections between patients with and without preoperative nasal MRSA colonization | Intervention period 2 years

SECONDARY OUTCOMES:
The incidence of MRSA infections between intervention and control period. | Intervention period 2 years, control period 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hyogo College of Medicine, Nishinomiya, Hyōgo, Japan